CLINICAL TRIAL: NCT02552836
Title: Evaluation of Two Psychotherapies for Depressed Patients With Parkinson's Disease
Brief Title: Efficacy of Psychotherapy for Depressed Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Montfort (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Montfort Hospital
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Depression; Parkinson's Disease
MeSH Terms: conditions — Depression; Parkinson Disease | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interpersonal Psychotherapy (IPT) (Experimental): Patients assigned to IPT will receive 12 sessions of individual therapy of approximately 50 minutes duration. Therapy will be manualized and slightly adapted to meet the needs of patients with Parkinson's Disease. Therapy focuses on one of four interpersonal events that are linked with onset or maintenance of depression (role transition, role disputes, unresolved grief, and interpersonal deficits).
  Interventions: Behavioral: Interpersonal Psychotherapy
- Supportive Psychotherapy (SP) (Active Comparator): Patients assigned to SP will receive 12 sessions of individual therapy of approximately 50 minutes duration. SP strives to create a supportive therapeutic relationship by emphasizing non-specific therapeutic interactions and techniques. Therapy will be manualized,
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy — A 12-week intervention that focuses on resolving interpersonal stressors that are linked to the onset, maintenance or exacerbation of depressive symptoms
  Arms: Interpersonal Psychotherapy (IPT)
Behavioral: Supportive Psychotherapy — A 12-week intervention that focuses on non-specific factors that contribute to therapy outcome
  Arms: Supportive Psychotherapy (SP)

SUMMARY:
The primary aim of this randomized controlled trial is to determine the acute antidepressant efficacy of interpersonal psychotherapy (IPT) in depressed patients with Parkinson's Disease.

DETAILED DESCRIPTION:
The primary aim of this study is to determine whether IPT is more efficacious than an intervention that controls for non-specific factors (i.e., supportive psychotherapy) in reducing depressive symptoms. A secondary aim is to determine whether IPT is better than supportive therapy in improving quality of life, interpersonal functioning, attachment patters, and motor symptoms, and whether treatment gains are durable at 6-months follow-up. An exploratory aim of the study is identify moderators and mediators of treatment outcome. Patients who meet study criteria will be randomly assigned to either 12 sessions of IPT or 12 sessions of supportive therapy. The primary efficacy measure (Hamilton Depression Rating Scale) will be administered at baseline, weeks 6 and 12, and at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with idiopathic Parkinson's disease and between stages 1 and 3 in the modified Hohn & Yahr Clinical Staging Scale
* Diagnosis of a depressive disorder
* Score ≥ 12 on the 17-item Hamilton Depression Rating Scale
* Living independently

Exclusion Criteria:

* History of bipolar disorder or psychotic symptoms (other than drug induced)
* Substance-related disorders in the last 12 months
* Acutely suicidal or history of suicide attempts in the past 5 years
* Presence of cognitive deficits (i.e., score ≤ 24 on the Mini Mental Status Exam) or history of significant cognitive disorders
* Presence of other significant neurological problems
* Presence of unstable comorbid medical conditions
* Currently receiving psychotherapy
* Unable to attend weekly therapy sessions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-A) | Change from baseline to week 12 and 6-months follow-up
  17-item clinician rated scale that assesses severity of depressive symptoms

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | Change from baseline to week 12 and 6-months follow-up
  The BDI is a self report measure of depressive symptoms
Beck Anxiety Inventory (BAI) | Change from baseline to week 12 and 6-months follow-up
  The BAI is a self-report measure of anxiety symptoms
Parkinson's Disease Questionnaire (PDQ-39) | Change from baseline to week 12 and 6-months follow-up
  Self-report questionnaire that assesses quality of life in patients with Parkinson's Disease
Interpersonal Relationships Inventory (IPRI) | Change from baseline to week 12 and 6-months follow-up
  Self-report inventory that measures aspects of interpersonal relationships
Experiences in Close Relationship Scale-Revised (ECR-R) | Change from baseline to week 12 and 6-months follow-up
  Self-report scale that assesses attachment style in adult relationships
Movement Disorders Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Change from baseline to week 12 and 6-months follow-up
  Clinician rated scale that provides comprehensive coverage of motor symptoms in Parkinson's Disease

CONTACTS AND LOCATIONS:
Overall Officials: Diana Koszycki, PhD, Principal Investigator — Montfort Hospital and the University of Ottawa
Locations (2):
- Canada (2):
  - The Ottawa Hospital and University of Ottawa, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No
No plan to share data